CLINICAL TRIAL: NCT03353441
Title: Effects of Microencapsulated Sublingual Glycine (Bidicin) on Cognitive Performance in Healthy Men After an Acute Stressor - a Randomized, Partly Double-blind Placebo-controlled Clinical Trial
Brief Title: Effects of Microencapsulated Sublingual Glycine (Bidicin) on Cognitive Performance in Healthy Men After an Acute Stressor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daacro (Network)
Collaborators: OOO MNPK BIOTIKI (Unknown)
Responsible Party: Principal Investigator, Juliane Hellhammer, PhD, Daacro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BI02-2017
Record Dates: First submitted 2017-11-10; First posted 2017-11-27 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Healthy; Stress, Psychological; Cognitive Impairment
Keywords: Verbal Learning and Memory Test (VLMT); Stroop Test; Attention; Working Memory; Learning and recognition; CogTrack
MeSH Terms: conditions — Stress, Psychological; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Partly double-blind (Glycine (MSG), Placebo, control without treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glycine (MSG) (Active Comparator): Microencapsulated Sublingual Glycine (MSG): 1 tablet prior to TSST; 1 tablet after the TSST
  Interventions: Dietary Supplement: Microencapsulated Sublingual Glycine (MSG)
- Placebo (Placebo Comparator): Lactose: 1 tablet prior to TSST; 1 tablet after the TSST
  Interventions: Dietary Supplement: Placebo
- No treatment (No Intervention)

INTERVENTIONS:
Dietary Supplement: Microencapsulated Sublingual Glycine (MSG) — Glycine (MSG) tablet
  Other Names: Bidicin
  Arms: Glycine (MSG)
Dietary Supplement: Placebo — Lactose tablet manufactured to mimic Glycine (MSG) tablet
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether intake of Glycine (MSG) leads to an increase of cognitive performance after an acute stressor compared to placebo. One group will receive verum, one group placebo and one group will not receive any intervention. Cognitive testing will be performed in connection with the Trier Social Stress Test (TSST).

DETAILED DESCRIPTION:
Stress can enhance or impair memory performances depending on the timing of the stressor and the timing of the memory processes in relation to the stressor. If stress occurs directly before or during the retrieval of information, the performance is impaired. Decreased performances using an acute stressor were also observed for other domains of cognitive functioning like working memory, interference control, cognitive flexibility and attention tasks.

Glycine, the simplest of the amino acids, is an essential component of important biological molecules, a key substance in many metabolic reactions, the major inhibitory neurotransmitter in the spinal cord and brain stem, and an anti-inflammatory, cytoprotective, and immune modulating substance. Studies have found positive effects of Glycine on episodic memory retrieval and in a word retrieval task.

To assess the effect of Glycine (MSG) on cognitive performance after an acute stressor, subjects perform baseline cognitive testing before intake of investigational products (Glycine (MSG), placebo or nothing) and participation in a stress test (Trier Social Stress Test - TSST). After the TSST stress-induced changes in cognitive performance are assessed. A second treatment intake takes place between the first and the remaining cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* subject signs the informed consent to participate in the study
* normally stressed subjects as verified by the TICS questionnaire with scores >3 and <37

Exclusion Criteria:

* smoker
* any known allergies to the test substances
* lactose intolerance
* any known addiction to drugs and/or alcohol
* hyper- or hypotension (except for those whose blood pressure is stable using medication for more than 3 months)
* known hyper- or hypothyroidism unless treated and under control (stable for more than 3 months)
* any known current/acute or chronic physical or psychological diseases besides minor medical conditions (e.g. seasonal allergies)
* intake of any medication which may affect the cognitive performance (e.g. psychotropics, sedating or stimulating medication)
* any color vision impairment (e.g. red-green deficiency)
* intake of dietary supplements or homoeopathic remedies during 2 weeks before V1 or during the study conduction
* consumption of alcohol during 2 days before V1 or during the study conduction
* excessive caffeine consumption (>400 mg caffeine/day or >= 4 cups of caffeinated coffee)
* on a strict diet or practicing sport, extensively
* attending an exam one week before and after the study participation
* subjects having previously participated in the TSST
* employee of the sponsor or Contract Research Organisation (CRO)
* Investigator doubts truthfulness of self-reported health information
* not suitable because of limited verbal and cognitive abilities

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Delayed memory performance after the TSST (correct words) | 20 minutes after second product intake
  Efficacy of the intake of Glycine (MSG) on performance in the Verbal Learning and Memory Test (VLMT) delayed recall task (number of correct words) compared to placebo and control group

SECONDARY OUTCOMES:
Delayed memory performance before and during the TSST | 15 minutes before and 42 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on performance in the Verbal Learning and Memory Test (VLMT) delayed recall task (number of correct words, number of perseverations and wrong words) compared to placebo and control group
Immediate memory performance before and after the TSST | 44 minutes before, 13 and 48 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on Performance in the Verbal Learning and Memory Test (VLMT) immediate recall task (number of correct words, decreased number of perseverations and wrong words) compared to placebo and control group
VAS stress | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute stress compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
VAS anxiety | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute anxiety compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
VAS insecurity | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute insecurity compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
VAS sleepiness | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute sleepiness compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
VAS tension | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute tension compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
VAS lack of energy | 20 minutes, 37 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on subjective evaluation of acute lack of energy compared to placebo and control group measured on a Visual Analogue Scale (VAS). The VAS is a 10cm bipolar visual scale ranging from "not at all" to "highly". VAS scores are obtained by using a ruler and measuring the position of the participant's mark with millimeter precision. To control for possible variations due to printing, the total length of the line is also measured and percentage scores for each subject are computed. Percentage scores range from 0-100.
STAI-state | 20 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on state anxiety as measured by the State Trait Anxiety Inventory (STAI) compared to placebo and control group. The STAI-state measures anxiety as a temporary emotional state and comprises 20 items. Answers are given on a four-point rating scale ranging from 1 = "not at all" to 4 = "very true". Some STAI questions relate to the absence of anxiety, and are reversely scored. For analysis of the STAI-scale, items are combined in one scale, which then informs about state anxiety. The score range is 20-80; higher scores indicate more anxiety.
Systolic and diastolic blood pressure | 25 minutes and 46 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on blood pressure in response to the TSST compared to placebo and control group
Delayed memory performance after the TSST (perseverations, wrong words) | 20 minutes after second product intake
  Efficacy of the intake of Glycine (MSG) on performance in the Verbal Learning and Memory Test (VLMT) delayed recall task (decreased number of perseverations and wrong words) compared to placebo and control group
Cognitive performance before and after the TSST (Stroop) | 10 minutes before first product intake and 23 minutes after second product intake
  Efficacy of the intake of Glycine (MSG) on performance in the Stroop test (speed and accuracy) compared to placebo and control group
Cognitive performance before and after the TSST (CogTrack) | 40 minutes before first product intake, immediately after second product intake
  Efficacy of the intake of Glycine (MSG) on performance in attention, working memory, learning and recognition tasks of CogTrack compared to placebo and control group
Heart rate | Continous measurement starting 10 minutes after first product intake and ending 10 minutes after second product intake
  Efficacy of the intake of Glycine (MSG) on heart rate in response to the TSST compared to placebo and control group
Salivary Cortisol | 45, 10 minutes before first product intake, 28, 46, 55 minutes after first product intake, 10, 20, 35 and 50 minutes after second product intake
  Efficacy of the intake of Glycine (MSG) on salivary cortisol raw values in response to the TSST compared to placebo and control group

OTHER OUTCOMES:
TICS | Baseline
  Do Trier Inventory for Chronic Stress (TICS) scores differ between groups? The TICS includes 57 items. Stress chronicity is measured by the frequency of stressful events perceived retrospectively within the last 3 months. Answers are given on a five-point rating scale, where 0 resembles "never" and 4 "very often". For analysis the questionnaire items are assigned to 10 scales: Work overload (range 0-32), Social overload (0-24), Pressure to succeed (0-36), Work dissatisfaction (0-32), excessive demands at work (0-24), Lack of social recognition (0-16), Social stress (0-24), Social isolation (0-24) and Chronic worrying (0-16); the last scale presents a Screening scale for chronic stress (0-48). Scores are obtained by summing up the values of the scale specific questionnaire items.
STAI-trait | Baseline
  Do State Trait Anxiety Inventory (STAI) trait scores differ between groups? The STAI-trait measures anxiety as a personality trait and comprises 20 items. Answers are given on a four-point rating scale ranging from 1 = "almost never" to 4 = "almost always". Some STAI questions relate to the absence of anxiety, and are reversely scored. For analysis of the STAI-scale, items are combined in one scale, which then informs about trait anxiety. The score range is 20-80; higher scores indicate more anxiety.
Mental arithmetic performance during the TSST | 37.5 minutes after first product intake
  Efficacy of the intake of Glycine (MSG) on arithmetic performance compared to placebo and control group. One part of the Trier Social Stress Test (TSST) is a mental arithmetic task. The subject is asked to stepwise subtract 17 from 2023 as quickly and correctly as possible. Performance will be measured by counting how many numbers the subject enumerates and how many times the subject has to restart. Furthermore, the lowest correct number and the shortest run will be recorded.
eCB levels | 45, 10 minutes before first product intake, 28, 46, 55 minutes after first product intake, 10, 20, 35 and 50 minutes after second product intake
  Exploration of endocannabinoid levels (eCB)
Blood Glucose levels | 75 minutes before first product intake, 25 and 46 minutes after first product intake
  Exploration of blood glucose levels

CONTACTS AND LOCATIONS:
Locations (1):
- daacro GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwabe L, Wolf OT. Stress and multiple memory systems: from 'thinking' to 'doing'. Trends Cogn Sci. 2013 Feb;17(2):60-8. doi: 10.1016/j.tics.2012.12.001. Epub 2013 Jan 2. PMID 23290054
- [Background] Shields GS, Sazma MA, McCullough AM, Yonelinas AP. The effects of acute stress on episodic memory: A meta-analysis and integrative review. Psychol Bull. 2017 Jun;143(6):636-675. doi: 10.1037/bul0000100. Epub 2017 Apr 3. PMID 28368148
- [Background] Shields GS, Sazma MA, Yonelinas AP. The effects of acute stress on core executive functions: A meta-analysis and comparison with cortisol. Neurosci Biobehav Rev. 2016 Sep;68:651-668. doi: 10.1016/j.neubiorev.2016.06.038. Epub 2016 Jun 28. PMID 27371161
- [Background] Lupien SJ, Gillin CJ, Hauger RL. Working memory is more sensitive than declarative memory to the acute effects of corticosteroids: a dose-response study in humans. Behav Neurosci. 1999 Jun;113(3):420-30. doi: 10.1037//0735-7044.113.3.420. PMID 10443770
- [Background] Olver JS, Pinney M, Maruff P, Norman TR. Impairments of spatial working memory and attention following acute psychosocial stress. Stress Health. 2015 Apr;31(2):115-23. doi: 10.1002/smi.2533. Epub 2014 Jan 3. PMID 24395182
- [Background] Schoofs D, Preuss D, Wolf OT. Psychosocial stress induces working memory impairments in an n-back paradigm. Psychoneuroendocrinology. 2008 Jun;33(5):643-53. doi: 10.1016/j.psyneuen.2008.02.004. Epub 2008 Mar 21. PMID 18359168
- [Background] Shields GS, Trainor BC, Lam JC, Yonelinas AP. Acute stress impairs cognitive flexibility in men, not women. Stress. 2016 Sep;19(5):542-6. doi: 10.1080/10253890.2016.1192603. Epub 2016 Jun 20. PMID 27230831
- [Background] Gundersen RY, Vaagenes P, Breivik T, Fonnum F, Opstad PK. Glycine--an important neurotransmitter and cytoprotective agent. Acta Anaesthesiol Scand. 2005 Sep;49(8):1108-16. doi: 10.1111/j.1399-6576.2005.00786.x. PMID 16095452
- [Background] File SE, Fluck E, Fernandes C. Beneficial effects of glycine (bioglycin) on memory and attention in young and middle-aged adults. J Clin Psychopharmacol. 1999 Dec;19(6):506-12. doi: 10.1097/00004714-199912000-00004. PMID 10587285
- [Background] Schwartz BL, Hashtroudi S, Herting RL, Handerson H, Deutsch SI. Glycine prodrug facilitates memory retrieval in humans. Neurology. 1991 Sep;41(9):1341-3. doi: 10.1212/wnl.41.9.1341. PMID 1653913
- See also: daacro homepage — http://www.daacro.de